CLINICAL TRIAL: NCT06348667
Title: Randomized, Controlled, Single-Blind, Longitudinal Experimental Study With Follow-up on the Effects of a Short- and Long-term 'Blackboard' Intervention on Ankle Stability and Mobility in Older Adults
Brief Title: Effects of a Short- and Long-term 'Blackboard' Intervention on Ankle Stability in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rodrigo Martín-San-Agustin, Assistant Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3184794
Record Dates: First submitted 2024-03-26; First posted 2024-04-05 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Fall
Keywords: Ankle stability; Ankle mobility; Balance training; Older Adults

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 16 subjects who will perform BB exercises twice a week for 5 weeks under the supervision of a physiotherapist.
  Each session (50') will include a warm-up of 10' of slow walking, joint mobility, and stretching. Then, BB exercises will be performed, followed by 10' of relaxation and stretching to cool down.
  BB exercises:
  * Ankle mobility: single-leg ankle dorsiflexion movements in a standing position on the BB with slight assistance from the parallel bars to perform the movement correctly. The BB will be set with the forefoot fixed and the rearfoot with medial drop, to facilitate dorsiflexion by combining dorsal flexion and pronation. 3 sets of 15 repetitions, with a 1' rest between sets.
  * Balance: BB will be set with instability in the forefoot and fixed rearfoot, to produce mediolateral instability of the CoP. The exercise will be maintaining balance on the BB while attempting to keep the lateral edges of the board from touching the ground. Five rounds of 40" work and 1' rest.
  Interventions: Other: Specific ankle stability exercises
- Control (Active Comparator): 16 participants who will perform their conventional exercises protocol. The group exercise sessions (45') take place twice a week. Participants sit in a circle in the room, with the physiotherapist in the center to provide instructions, and perform:
  * Warm-up: 5' of joint mobility exercises. Shoulder rotations, elbow flexion and extension, knee flexion and extension, ankle rotations, and standing up and sitting down 5 times.
  * Main part: 25-30' (with music). Energetic arm movements, e.g. raising and lowering, front and back, inward and outward arm circles, and lateral shoulder raises like "little birds"... These exercises are performed fast within a controlled ROM. CORE work is done while seated on the edge of the chair, bringing knees to the shoulders and moving the legs up and down. Finally, they stand up and sit down several times, and try to maintain an isometric squat position.
  * Cool down: 5-7' of stretching, mainly consisting of active neck mobility and arm stretching.
  Interventions: Other: Conventional physiotherapy exercises program

INTERVENTIONS:
Other: Specific ankle stability exercises — Exercise program specifically designed to address ankle dorsiflexion and mediolateral displacement of the center of pressure, using the described device (BB). Done twice a week for 5 weeks.
  Arms: Experimental
Other: Conventional physiotherapy exercises program — Conventional exercise program performed in the center twice a week, of which all participants are part.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of adding specific Blackboard Training (BB) exercises to conventional physiotherapy in improving foot and ankle parameters essential for fall prevention among older adults.

The main questions it aims to answer are:

1. Can the addition of BB exercises improve ankle dorsiflexion mobility?
2. Can the addition of BB exercises enhance single-leg stability and control of mediolateral displacement of the center of pressure?

Participants will be divided into control and intervention groups. Both groups will receive their usual conventional physiotherapy exercises. The intervention group will undergo a 5-week program comprising 10 sessions of BB exercises targeting ankle mobility and balance.

Participants will be asked to:

* Perform 3 sets of 15 repetitions for assisted ankle dorsiflexion mobility.
* Engage in 5 rounds of 40-second balance exercises using the BB.

Researchers will compare the intervention group's outcomes with those of the control group to determine the effectiveness of adding BB exercises in improving foot and ankle parameters related to fall prevention.

DETAILED DESCRIPTION:
Age serves as a predictor of single-leg stability, ankle dorsiflexion range, and plantar flexor strength loss in older adults. Various factors contribute to their heightened risk of falls, such as foot pain, reduced ankle and big toe mobility, increased pressure on specific foot regions during stance, and greater mediolateral displacement of center of pressure.

Exercise interventions have strong support in the field of fall prevention. In turn, foot flexor muscle fatigue has been associated with increased displacement of the center of pressures, so training of this muscles may be useful. While several fall prevention strategies for older adults have shown positive outcomes, some studies face limitations like small sample sizes or insufficient improvement in static balance, possibly due to low exercise intensity and specificity.

The conventional use of instability devices like the BOSU, Wobble board, Airex, or Swiss ball presents challenges in older adult contexts due to their bulkiness and indiscriminate instability. Hence, a specific instability training approach could be interesting to address fall risk factors.

This study proposes a Blackboard Training (BB) exercise intervention for older adults, known for its portability, small size, and adaptability, comparable in effectiveness to traditional devices like the BOSU or Wobble board in activating Peroneus longus muscle, essential for single-leg stability.

Participants will be divided into control and intervention groups, both receiving their usual conventional physiotherapy exercises. The intervention group will undergo a 5-week program comprising 10 sessions. Measurements will be taken pre-study, one week prior, post-study completion, and at a follow-up one month later to assess the duration of observed changes. Each session, lasting 50 minutes, will include a warm-up, BB exercises targeting ankle mobility and balance, and a cool-down. Safety precautions, such as parallel bars for support, will be provided during balance exercises. Specific BB exercises will be: 3 sets of 15 repetitions for assisted ankle dorsiflexion mobility and 5 rounds of 40-second balance exercises.

The analyzed variables will include ankle and big toe range of motion (ROM), the Lunge test, bipedal and monopodal stabilometry, strength of ankle and foot, the Timed-Up-and-Go test and the Single-leg Stance Test.

The hypothesis is that adding specific BB training to conventional physiotherapy for older adults can improve foot and ankle parameters essential for fall prevention, including ankle dorsiflexion and single-leg support. Improvement in ankle dorsiflexion and better control of mediolateral displacement of the center of pressure are expected outcomes.

ELIGIBILITY:
Inclusion criteria:

* Ability to walk at least 5 meters without the need for technical aids
* Achieving a minimum score of 24 on the Mini-Mental State Examination, ensuring cognitive capacity to understand the study
* Attaining a minimum score of 19 on the Tinetti scale

Exclusion criteria:

* Not having participated in any specific stability or ankle training program in the last 6 months
* Not experiencing any musculoskeletal or neural disorders that could hinder study participation (e.g., diabetic foot, hemiplegia, or amputations)
* Individuals at severe risk of falling and those who are solely able to stand without being able to walk, according to the Tinetti scale

Ages: 75 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Foot and ankle pain | Pre, after 5 weeks of intervention, after 1 month of the end of the study
  Foot-Function Index (FFI) scale. The FFI consists of 23 items divided into 3 subscales that quantify the impact of foot pathology on pain, disability, and activity limitation. It offers a score from 0 to 267, with higher scores indicating worse outcomes. The total score obtained on the scale is divided by 207 and multiplied by 100 to obtain a final percentage.
Foot and ankle strength | Pre, after 5 weeks of intervention, after 1 month of the end of the study
  Suiff Pro dynamometer. Movements: dorsal and plantar flexion, inversion, eversion of the ankle. Flexion and extension of the big toe.
Foot and ankle ROM | Pre, after 5 weeks of intervention, after 1 month of the end of the study
  Video recording + Kinovea. Movements: dorsal and plantar flexion, inversion, eversion of the ankle. Flexion and extension of the big toe.
Ankle dorsiflexion under load | Pre, after 5 weeks of intervention, after 1 month of the end of the study
  Weight bearing Lunge test. This test is used to assess ankle dorsiflexion. The movement will be recorded for later processing with Kinovea to determine the angle.
Center of pressures variations (anteroposterior and mediolateral center of pressure displacement, velocity, and total surface) | Pre, after 5 weeks of intervention, after 1 month of the end of the study
  K-Force plates will be used during bipedal and monopodal stances. First on a firm surface with eyes open, and then with eyes closed. The same procedure will be performed on a soft surface.
Monopodal stability | Pre, after 5 weeks of intervention, after 1 month of the end of the study
  Single-leg Stance Test. During this test, the time that the participant is able to maintain single-leg stance without arm support and with eyes open is recorded.
Functional stability | Pre, after 5 weeks of intervention, after 1 month of the end of the study
  Timed Up and Go test. In this test, the participant is seated in a chair with a cone placed 3 meters in front of them. Upon signal, they stand up, walk to the cone, walk around it, come back, and sit down again. The time taken to complete the task will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Martín-San Agustín, Doctor, Principal Investigator — University of Valencia
Locations (1):
- Rodrigo Martin-San Agustin, Valencia, Spain